CLINICAL TRIAL: NCT05579886
Title: Evaluating the Success of Refitting Lens Wearers With MyDay Multifocal, Who Are Already Adapted to Clariti 1Day Multifocal 2-Add Design
Brief Title: Evaluating Two Multifocal Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EX-MKTG-140
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lens (Active Comparator): All participants wore the Control Lens for 2 weeks (Period 1)
  Interventions: Device: Control Lens
- Test Lens (Experimental): All participants wore the Test Lens for 2 weeks (Period 2)
  Interventions: Device: Test Lens

INTERVENTIONS:
Device: Control Lens — Daily disposable multifocal soft lens with 2 add design (2ADD) for 2 weeks
  Arms: Control Lens
Device: Test Lens — Daily disposable multifocal soft lens with 3 add design (3ADD) for 2 weeks
  Arms: Test Lens

SUMMARY:
The objective of the study was to adapt existing multifocal soft lens wearers to a Control Lens for at least 2 weeks and then evaluate the success of switching them to the Test Lens, with a review after 2 weeks.

DETAILED DESCRIPTION:
This prospective, bilateral eye, open label, non-randomized study compared the performance of 2 different designs of daily disposable multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

A person was eligible for inclusion in the study if he/she:

1. Was at least 42 years of age and had full legal capacity to volunteer;
2. Had read and signed an information consent letter;
3. Self-reported having had a full eye examination in the previous two years;
4. Anticipated being able to wear the study lenses for at least 8 hours a day, 5 days a week;
5. Was willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wore multifocal soft contact lenses, for the past 3 months minimum (NOTE: the habitual contact lens type was restricted such that no more than one third were to be the clariti 1 day multifocal and no more than one third were to be MyDay multifocal (this included their equivalent private label brand name);
7. Had refractive astigmatism no higher than -0.75DC in each eye;
8. Was presbyopic and required a reading addition of at least +0.75D and no more than +2.50D in each eye;
9. Could be fit and achieved binocular distance vision of at least 20/30 Snellen (or +0.20 logMAR) which participants also deemed to be 'acceptable', with the available study lens parameters (powers +4.00 to -6.00DS)

Exclusion Criteria:

A person was excluded from the study if he/she:

1. Was participating in any concurrent clinical or research study;
2. Had any known active ocular disease and/or infection that contraindicated contact lens wear;
3. Had a systemic condition that in the opinion of the investigator may have affected a study outcome variable;
4. Was using any systemic or topical medications that in the opinion of the investigator may have affected contact lens wear or a study outcome variable;
5. Had known sensitivity to the diagnostic sodium fluorescein to be used in the study;
6. Self-reported as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Had undergone refractive error surgery or interocular surgery.

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sacco, Principal Investigator — Sacco Eye Group; Shane Kannarr, Principal Investigator — Kannarr Eye Care; Katherine Bickle, Principal Investigator — ProCare Vision Center; Michael Cymbor, Principal Investigator — Nittany Eye Associates; Roxanne Achong-Coan, Principal Investigator — Coan Eye Care & Optical Boutique
Locations (5):
- United States (5):
  - Coan Eye Care & Optical Boutique, Ocoee, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Center, Granville, Ohio
  - Nittany Eye Associates, State College, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Lens (2ADD): All participants wore the Control Lens for 2 weeks (Period 1)
- Test Lens (3ADD): All participants wore the Test Lens for 2 weeks (Period 2)
Period: Period 1: Control Lens, 2 Weeks
Arm/Group | Control Lens (2ADD) | Test Lens (3ADD)
Started | 60 | 0 (All participants received Control Lens in Period 1.)
Completed | 60 | 0
Not Completed | 0 | 0
Period: Period 2: Test Lens, 2 Weeks
Arm/Group | Control Lens (2ADD) | Test Lens (3ADD)
Started | 0 (All participants received Test Lens in Period 2.) | 60
Completed | 0 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Comfort Just After Lens Insertion
Description: Subjective rating measured on a scale of 0-10, 0.5 steps, where 0=Painful, 10=Can't feel the lenses.
Time Frame: 2 weeks
Population: All participants wore Control Lens and Test Lens in sequential order.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Lens (2ADD): Participants that received Control Lens
- Test Lens (3ADD): Participants that received Test Lens
Arm/Group | Control Lens (2ADD) | Test Lens (3ADD)
Number analyzed (Participants) | 60 | 60
score on a scale | 9.1 (1.4) | 9.2 (1.1)

ADVERSE EVENTS:
Time Frame: From dispense to study exit, approximately 6-8 weeks.
Arm/Group | Control Lens (2ADD) | Test Lens (3ADD)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 1/60 | 0/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Lens (2ADD) (N=60) | Test Lens (3ADD) (N=60)
Influenza (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT05579886/Prot_SAP_000.pdf